CLINICAL TRIAL: NCT03727360
Title: Exercise for Brain Health in the Fight Against Alzheimer's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, College Park (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Johns Hopkins University (Other); Marquette University (Other); University of Maryland, Baltimore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 1115946; 1R01AG057552 (NIH)
Record Dates: First submitted 2018-10-26; First posted 2018-11-01 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Healthy Cognition
Keywords: Walking Exercise; Flexibility Exercise; Cognition; Memory; Magnetic Resonance Imaging
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants and outcomes assessors are masked to APOE genotype. We do not share any data with care providers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Training (Experimental): Group exercise and treadmill walking
  Interventions: Other: Exercise Training
- Flexibility Control (Active Comparator): Group exercise and flexibility exercise
  Interventions: Other: Flexibility Control

INTERVENTIONS:
Other: Exercise Training — Supervised exercise conducted four days per week for six months.
  Arms: Exercise Training
Other: Flexibility Control — Supervised exercise conducted four days per week for six months.
  Arms: Flexibility Control

SUMMARY:
The investigators aim to compare the effects of a 6-month moderate intensity exercise training (ET) intervention to a low intensity flexibility exercise control condition (FC) on brain function, cognition, and physical function in cognitively healthy and physically inactive older adults (ages 60-80). Apolipoprotein E epsilon4 (APOE-ε4) allele carriers are known to be at substantially greater risk for cognitive decline and Alzheimer's disease (AD). Cognitively intact APOE-ε4 allele carriers, and non-carriers, will be randomly assigned to 6-months of either supervised moderate intensity aerobic exercise training (ET) or supervised flexibility exercise control (FC). The ET and FC each contain a group based exercise component and are run in local retirement communities near College Park, MD, or on the University of Maryland College Park campus. The primary aims of the study are to compare pre-intervention to post-intervention changes in episodic memory performance and MRI biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* 60 to 80 years old
* Fluent in English
* Willingness to make the time commitment to participate in the project, including randomization to treatments
* Physically inactive (physical activity not more than 2 days per week for the past 6 months)
* Physician consent to undergo an exercise stress test and engage in moderate intensity exercise
* Determined to be safe for MRI

Exclusion Criteria:

* Neurological illnesses/conditions such as cerebral palsy, epi¬lepsy, brain tumor, chronic meningitis, multiple scle¬rosis, pernicious anemia, normal-pressure hydrocephalus, HIV infection, Parkinson's disease, and Huntington's disease
* Untreated hypertension, glaucoma, and chronic obstructive pul¬monary disease
* Untreated severe major depression
* Substance abuse or dependence
* Current use of psychoactive medications, except selective serotonin/norepinephrine reuptake inhibitor antidepressants
* Use of acetylcholinesterase inhibitors (e.g., Aricept)
* Unstable or severe cardiovascular disease or asthmatic condition
* History of transient ischemic attack, cerebral ischemia, or clinically diagnosed stroke
* Diagnosis of mild cognitive impairment or dementia, or objective evidence of cognitive impairment

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2018-10-08 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline to 6 months in Rey Auditory Verbal Learning Test Sum of Trials 1-5 | Baseline and 6 months
Change from Baseline to 6 months in Resting Cerebral Blood Flow | Baseline and 6 months

SECONDARY OUTCOMES:
Change from Baseline to 6 months in VO2peak | Baseline and 6 months
  Estimated peak rate of oxygen consumption, a measure of cardiorespiratory fitness
Change from Baseline to 6 months in 6 Minute Walk Test | Baseline and 6 months
  Distance walked in 6 minutes

CONTACTS AND LOCATIONS:
Overall Officials: J. Carson Smith, PhD, Principal Investigator — University of Maryland
Locations (1):
- University of Maryland, Department of Kinesiology, College Park, Maryland, United States